CLINICAL TRIAL: NCT02071524
Title: Evaluation of the Effects of Fluid Therapy on Respiratory Mechanics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Università degli Studi di Ferrara (Other)
Responsible Party: Principal Investigator, Savino Spadaro, Researcher, Università degli Studi di Ferrara
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 22012014
Record Dates: First submitted 2014-01-28; First posted 2014-02-26 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Mechanical Ventilation Complication; Actual Impaired Fluid Volume

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cristalloid (Active Comparator): group cristalloid (ringer lactate)
  Interventions: Drug: Cristalloid administration
- colloids (Active Comparator): colloid: cristalloid in according to cardiac output
  Interventions: Drug: Group Colloid

INTERVENTIONS:
Drug: Group Colloid — Group Colloid: cristalloid 1:2 (gelofusine: ringer lactate)
  Arms: colloids
Drug: Cristalloid administration — Only Ringer Lactate administration
  Arms: Cristalloid

SUMMARY:
The investigators hypothesize that large doses of fluids used during intraoperative could affect lung parenchyma structure and, consequently, gas exchange and respiratory mechanics. The purpose of this study is to evaluate fluids effects on oxygenation, respiratory mechanics, by using two different solutions: crystalloid or colloid.

DETAILED DESCRIPTION:
Inclusion Criteria:

* patients undergoing elective abdominal, thoracic, vascular surgery
* minimum age 18 years
* informed consent

Exclusion Criteria:

* patients with severe cardiomyopathy or severe heart failure
* history of coagulation disorders
* patients with severe cardiovascular or respiratory disorders
* renal insufficiency

Respiratory mechanic parameters (i.e., inspiratory peak pressure, plateau pressure, total airway resistance, and static compliance) are obtained .Blood samples are drawn simultaneously from the arterial catheters for gas analysis. Data were collected after induction of anesthesia (T0) after 1 h (T1), 2 h (T2), 3 h (T3) and at the end of surgery.

Primary outcome: evaluate the fluids effects on oxygenation, respiratory mechanics

Secondary outcome: Incidence of surgery related complications

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective abdominal, thoracic, vascular surgery
* minimum age 18 years
* informed consent

Exclusion Criteria:

* patients with severe cardiomyopathy or severe heart failure
* history of coagulation disorders
* patients with severe cardiovascular or respiratory disorders
* renal insufficiency
* severe liver diseases

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-09; Primary Completion 2017-03 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
effects on oxygenation, respiratory mechanics | every 30 minutes till the end of surgery
  Lung compliance (l/cmH20), Airaway resistance (cmH2O/L/sec) and PaO2 will be measured

SECONDARY OUTCOMES:
Incidence of respiratory complications | 28 days
  Complications like acute respiratory failure, pneumonia and ARDS will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ferrara, Ferrara, Italy